CLINICAL TRIAL: NCT01696500
Title: NPB-01(Intravenous Immunoglobulin) Therapy for Patients With Stevens-Johnson Syndrome/ Toxic Epidermal Necrolysis Unresponsive to Corticosteroids.
Brief Title: Phase III Clinical Trial of NPB-01 in Patients With Stevens-Johnson Syndrome/ Toxic Epidermal Necrolysis Unresponsive to Corticosteroids.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPB-01-07/C-01
Record Dates: First submitted 2012-09-20; First posted 2012-10-01 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2013-10

CONDITIONS: Stevens-Johnson Syndrome; Toxic Epidermal Necrolysis
Keywords: IVIG in Stevens-Johnson syndrome; Toxic Epidermal Necrolysis; Patients with Stevens-Johnson syndrome; Toxic Epidermal Necrolysis unresponsive to corticosteroids
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPB-01 (Experimental)
  Interventions: Drug: Intravenous immunoglobulin

INTERVENTIONS:
Drug: Intravenous immunoglobulin

SUMMARY:
Patients diagnosed with Stevens-Johnson syndrome and Toxic Epidermal Necrolysis were confirmed based on the investigators national diagnostic criteria. Patients who meet all inclusion criteria and do not conflict with the exclusion criteria will receive NPB-01 (intravenous immunoglobulin) 400mg/kg/day for five consecutive days. Subsequently, efficacy of NPB-01 for therapy of Stevens-Johnson syndrome and Toxic Epidermal Necrolysis will be evaluated the disease evaluation score et al.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by 20 days after the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who the disease evaluation score is more than 14 at study medication received.
2. Patients with corticosteroids over 20mg/day(Prednisolone) at study medication received and continued this treatment more than 2 days.
3. Patients with treatment effect is insufficiency before study medication received and need additional treatment.
4. Patients aged more than twenty years old at informed consent.

Exclusion Criteria:

1. Patients who the SCORTEN score is more than 4 at study medication received.
2. Patients with multiple organ failure at study medication received.
3. Patients with severe respiratory disorder at study medication received.
4. Patients with Drug-induced hypersensitivity syndrome (DIHS) at informed consent.
5. Patients with malignancy during treatment at informed consent.
6. Patients treated with corticosteroids dosage is change at 2 days before study medication received.
7. Patients treated with corticosteroids pulse therapy(including semi-pulse therapy) at 2 days before study medication received.
8. Patients treated with plasmapheresis at 2 days before study medication received.
9. Patients treated with high-dose intravenous immunoglobulin at 28 days before informed consent.
10. Patients with history of shock or hypersensitivity for NPB-01.
11. Patients with IgA deficiency.
12. Patients with severe impaired liver function diagnosed virus hepatitis or cirrhosis et al.
13. Patients with more than 2mg/dL serum creatinine.
14. Patients with severe cerebro- or cardiovascular disorders.
15. Patients with high risk of thromboembolism.
16. Patients with hemolytic/hemorrhagic anemia.
17. Patients with severe decreased cardiac function.
18. Patients with decreased platelet less than 75,000/μL..

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
disease evaluation score | 7 days

SECONDARY OUTCOMES:
disease evaluation score | 4 ,10 ,20 days
avulsed skin area | 20 days
erythematous area | 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon Pharmaceutical Co., Ltd, Tokyo, Japan